CLINICAL TRIAL: NCT05422105
Title: Multicenter Evaluation of Diagnostic Performance of [18F]FPSMA-1007 PET/CT in Patients With Suspected Prostate Cancer
Brief Title: Diagnostic Performance of 18F-PSMA-1007 PET/CT in Suspected Prostate Cancer Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Primo Biotechnology Co., Ltd (Industry)
Collaborators: ABX advanced biochemical compounds GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: PB01-MCTNSPC
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Prostate Cancer; Prostate Neoplasm
Keywords: Prostate cancer; [18F]FPSMA-1007; mpMRI
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected Prostate Cancer
  Interventions: Drug: 18F-PSMA-1007

INTERVENTIONS:
Drug: 18F-PSMA-1007 — 18F-PSMA-1007 PET/CT
  Other Names: [18F]FPSMA-1007

SUMMARY:
The diagnostic tools for detecting patients with early prostate cancer are limited due to poor diagnostic performance. The positron emission tomography (PET) combination with the diagnostic radiopharmacy is a non-invasive tool to provide the molecular imaging of the whole body and offer more comprehensive physiological information and then can raise the diagnostic performance. Prostate-specific membrane antigen (PSMA)-targeting pharmaceuticals have been regarded as the most promising diagnostic tool to diagnose patients with prostate cancer. Currently, the 18F-PSMA-1007 as PSMA-targeting 18F-radiolabeled pharmaceuticals have developed and successfully used in patients with intermittent- and high-risk prostate cancer or recurrent prostate cancer. The study aims to understand the diagnostic performance of 18F-PSMA-1007 PET/CT in different-stage prostate cancer patients by initiating the first multicenter clinical trial of 18F-PSMA-1007 in Taiwan.

ELIGIBILITY:
Inclusion Criteria

1. The participants are male adults over 20 years old.
2. The participants are suspected prostate cancer patients by a serum PSA value of 4-20 ng/ml or a serum PSA value of < 4ng/ml but noted abnormal lesion by DRE.
3. The participants agree to receive TRUS Bx or mpMRI fusion Bx examination.
4. The participants are the first time to receive a prostatic biopsy.

Exclusion Criteria

1. The participants are diagnosed with prostate cancer before this study.
2. The participants have received any related treatment for prostate cancer.
3. The participants have chronic prostatitis.
4. The participants' serum hemoglobin lowers than 10 mg/dl within 1 month.
5. The participants' serum platelet lowers than 15 103/uL within 1 month.
6. The participants' serum prothrombin time (PT) is prolonged longer than 1.2-fold within 1 month.
7. The participants' serum active partial prothrombin time (aPPT) is prolonged longer than 45 seconds within 1 month.
8. The participants have hemorrhagic disease such as Hemophilia, Von Willebrand disease, thrombocytopenia, systemic Lupus Erythematosus, etc. within 6 months.
9. The participants have conditions of poor immunity status such as HIV infection, receiving treatment for other cancer, DM poor control, use of immunomodulator (ex.

   steroid, etc.) within 6 months.
10. The participants have hypertension poor control that is BP cannot be controlled lower than 140/90mmHg whether or not taking medication within 6 months.
11. The participants have suffered from CVA including infarctions and hemorrhages within 6 months.
12. The participants have suffered from angina including stable and unstable types within 6 months.
13. The participants have suffered from arrythmia poor control within 6 months.
14. The participants have suffered from liver dysfunction such as AST/ALT ratio >2、total bilirubin >1.5 mg/dL within 6 months.
15. The participants are allergic to any radiopharmaceutical or imaging agent.
16. The participants suffered stage IV chronic kidney disease (eGFR<30 mL/min/1.73 m2) within 6 months
17. The participants suffered acute kidney injury within 6 months.
18. The participants are absolute and relative contraindications to MRI examination.

Ages: 20 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with suspected prostate cancer had a serum PSA value between 4 and 20 ng/ml or a serum PSA value of < 4ng/ml but noted abnormal lesions by digital rectal examination.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Performance | 7-14 days after PET/CT
  Sensitivity, Specificity, NPV, PPV

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Tungs'Taichung Metro Harbor Hospital, Taichung
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided